CLINICAL TRIAL: NCT05901142
Title: The Feasibility of a Multi-phasic Exercise-based Intervention Utilising the Health Action Process Approach, Dyadic Coping and Wearable Technology in Women Before and After Surgery for Breast Cancer
Brief Title: Prehabilitation and RecOVERy From Surgery for Breast Cancer Study
Acronym: PROVERB
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospitals of Derby and Burton NHS Foundation Trust (Other)
Collaborators: University of Wolverhampton (Other); University of Hull (Other); Sheffield Teaching Hospitals NHS Foundation Trust (Other); University of Bath (Other); Aston University (Other); Staffordshire University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PROVERB
Record Dates: First submitted 2023-05-02; First posted 2023-06-13 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2024-08

CONDITIONS: Exercise; Breast Neoplasm Female
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Exercise-based multi-phasic, multi-modal intervention (Experimental): An exercise-based multi-phasic (pre-surgery and post-surgery) and multi-modal (exercise, targeted physiotherapy, dietary advice, and psychological coping and behaviour change) intervention
  Interventions: Behavioral: Exercise-based multi-phasic, multi-modal intervention

INTERVENTIONS:
Behavioral: Exercise-based multi-phasic, multi-modal intervention — Pre-op: 2*60min supervised; 1*30min unsupervised walking sessions per week Supervised session: Aerobic: 8*60secs star jump, squat thrust, high knees with 90sec rest. Elastic resistance: 2*10-12reps of chest press, seated row, leg press, 'lat' pulldown, and either abdominal flexion or lumbar extension-alternated, with 60-90sec rest. Targeted physiotherapy: general breathing exercises, active-assisted range of motion (RoM) exercises, and active-resisted RoM exercises
  Postop: 1*60min supervised exercise; unsupervised walking [2*30min weeks 1-2; 3*30min week 3; 4*30min weeks 4-6] session per week Supervised session: Aerobic: As above using full body extension, squat jump, static sprint in week 1-4. Progressed to those performed preoperatively from week 5. Elastic resistance: As above from week 4, performed 3*week. Targeted physiotherapy: As above, with active-assisted RoM progressing from 1*10reps in week 1, to 2*10reps in weeks 2-4, and 3*10reps in weeks 4-6

SUMMARY:
Background and study aims:

Nine out of ten women experience some negative effects due to their disease or its treatment such as anxiety, depression, weight gain and low quality of life. Research shows that exercise may help women overcome some of these effects. The investigators also know that most women become physically inactive after cancer treatment. Therefore, The investigators feel it is important that women get into a routine of doing regular exercise before they start their cancer treatment, this is called prehabilitation. The investigators believe that prehabilitation might help to build confidence and help women to continue exercising after their cancer treatment.

The investigators are doing this study to find out if a remote (NHS Attend Anywhere), multimodal (aerobic, resistance and targeted exercise), behavioural change (Health Action Process Approach (HAPA), dyadic coping (the collective effort to dealing with the stress of breast cancer diagnosis and treatment), and wearable technology), multiphasic (pre- and post-surgery) intervention is feasible in the short time frame between diagnosis of breast cancer and surgery (less than 31 days). The investigators would also like to find out whether it is feasible for women to begin an exercise rehabilitation programme two weeks after their operation. If successful, the results will potentially enable us in the future to tailor the support gievn to women to help them prepare and recover from breast cancer treatment.

ELIGIBILITY:
Inclusion Criteria:

* Females aged 18 years or older
* Scheduled to undergo elective surgery for biopsy-proven breast cancer (lumpectomy or mastectomy) for resection and/or reconstruction purposes
* Patients scheduled after diagnosis of invasive breast cancer and ductal carcinoma in situ (DCIS)
* Able to communicate in English and able to provide and understand informed consent
* Willing to participate in supervised and home-based exercise
* Have the approval of operating surgeon
* At least 2 weeks until surgery
* Access to a computer or smart device connected to the world wide web

Exclusion Criteria:

* Evidence in the medical record of an absolute contraindication for exercise [e.g., Heart insufficiency > New York Heart Association (NYHA) III or uncertain arrhythmia; uncontrolled hypertension; severe renal dysfunction (Estimated Glomerular Filtration Rate (eGFR) < 30%, Creatinine> 3 mg/dl); insufficient haematological capacity like either haemoglobin value below 8 g/dl or thrombocytes below 30.000/µL; reduced standing or walking ability].
* Metastatic breast cancer
* Current smokers
* Not fluent in written and spoken English
* Engaging in regular exercise (at least 150 min per week of moderate exercise or at least 75 min per week of vigorous exercise, or an equivalent combination of moderate and vigorous exercise). This criterion will be assessed via the Physical Activity Vital Signs (PAVS) questionnaire, which asks the following two questions: 1) "Please describe your level of physical activity, [first by] minutes per day, [followed by] number of days each week", and 2) "At what intensity (how hard): light (like a casual walk), moderate (like a brisk walk), or vigorous (like a jog/run)?" (Ball et al., 2016). The questionnaire is scored by multiplying the days by minutes of physical activity to create an estimate of minutes per week of at least moderate-to-vigorous physical activity.
* Symptoms of long-covid/post covid syndrome

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Estimated)
Dates: Start 2023-06-16 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Number of participants recruited during the 36 week recruitment period | Assessed immediately after the 36 week recruitment period
  The investigators aim to recruit 34 participants in 36 weeks, equating to a recruitment rate of approximately one patient each week.
Number of participants retained during the interventional period | Assessed 2 weeks post-surgery (T1), and immediately after the 6-weeks of postoperative exercise (T2)
  The investigators aim to retain 75% (n = 25) of our sample throughout the interventional period, which includes a perioperative (~4 weeks) and post operative multimodal intervention (~6 weeks)
Number of participants who completed at least 70% of supervised sessions and not lower than 60% for of unsupervised sessions, spanning both the pre- and postoperative periods. | Assessed 2 weeks post-surgery (T1), and immediately after the 6-weeks of postoperative exercise (T2)
  Adherence to remotely supervised exercise sessions (spanning both pre- and postoperative phases) is at least 70%, and not lower than 60% for adherence to unsupervised exercise sessions.
Number of participants who had an average daily wear time is ≥10 hours per day and ≥4 days per week | Assessed 2 weeks post-surgery (T1), and immediately after the 6-weeks of postoperative exercise (T2)
  Feasibility of using wearable technology in patients with cancer will be supported if daily wear time is ≥10 hours per day and ≥4 days per week
Number of participants who experienced adverse events during exercise testing, supervised exercise, or unsupervised exercise. | Assessed 2 weeks post-surgery (T1), immediately after the 6-weeks of postoperative exercise (T2), and immediately after the 3 months follow up post exercise period (T3)
  Safety of physical activity will be assessed by recording the number of adverse events occurring during exercise testing, remotely supervised exercise training, and unsupervised exercise training. Adverse events will be recorded on a standardised data collection form

SECONDARY OUTCOMES:
Change from baseline in Health Action Process Approach (HAPA) after preoperative intervention and surgery, 6 weeks postoperative intervention, and after a three month observational period | Assessed at baseline (T0), within 1 week of completing the 2 weeks post-surgery (T1), within 1 week of completing the 6-weeks of postoperative exercise (T2), and within 1 week of completing the 3-months follow-up post-exercise (T3)
  HAPA variables measuring beliefs and attitudes will be adapted from the 4-point response scale (1 completely false; 2 sometimes false; 3 sometimes true and 4 completely true).
Change from baseline in Dyadic coping after preoperative intervention and surgery, 6 weeks postoperative intervention, and after a three month observational period | Assessed at baseline (T0), within 1 week of completing the 2 weeks post-surgery (T1), within 1 week of completing the 6-weeks of postoperative exercise (T2), and within 1 week of completing the 3-months follow-up post-exercise (T3)
  The dyadic coping inventory assesses perceived stress communication and dyadic coping. The 37-item dyadic coping inventory includes several subscales not relevant to this study. As such, to alleviate participant burden only the following subscales will be considered;
  * Supportive dyadic coping of the partner (SDCP: items 5, 6, 8, 9, and 13)
  * Delegated dyadic coping of the partner (DDCP: items 12 and 14)
  * Common dyadic coping (CDC: items 31, 32, 33, 34, and 35)
  * Evaluation of dyadic coping (EDC: items 36) Participants rate each of these 13 items on a 5-point Likert scale (1 = very rarely to 5 = very often). Mean scores for individual subscales will be used in the analysis.
Change from baseline in European Organization for Research and Treatment of Cancer (EORTC) Breast Cancer-Specific Quality of Life (QLQ-BR23) after preoperative intervention and surgery, 6 weeks postoperative intervention, and a 3 month observation | Assessed at baseline (T0), within 1 week of completing the 2 weeks post-surgery (T1), within 1 week of completing the 6-weeks of postoperative exercise (T2), and within 1 week of completing the 3-months follow-up post-exercise (T3)
  Specific breast cancer-related symptoms will be assessed with the validated 23-item European Organization for Research and Treatment of Cancer (EORTC) Breast Cancer-Specific Quality of Life Questionnaire (QLQ-BR23). All of the scales and single-item measures range in score from 0 to 100. A high scale score represents a higher response level.
Change from baseline in European Organization for Research and Treatment of Cancer (EORTC) after preoperative intervention and surgery, 6 weeks postoperative intervention, and after a three month observational period | Assessed at baseline (T0), within 1 week of completing the 2 weeks post-surgery (T1), within 1 week of completing the 6-weeks of postoperative exercise (T2), and within 1 week of completing the 3-months follow-up post-exercise (T3)
  In concordance with the International Consortium for Health Outcomes Measurement, quality of life will be assessed with the validated 30-item self-assessment questionnaire of the European Organization for Research and Treatment of Cancer (EORTC QLQ-C30). All of the scales and single-item measures range in score from 0 to 100. A high scale score represents a higher response level.
Change from baseline in BREAST-Q-Satisfaction after preoperative intervention and surgery, 6 weeks postoperative intervention, and after a three month observational period | Assessed at baseline (T0), within 1 week of completing the 2 weeks post-surgery (T1), within 1 week of completing the 6-weeks of postoperative exercise (T2), and within 1 week of completing the 3-months follow-up post-exercise (T3)
  Satisfaction with breast(s) will be assessed via BREAST-Q-Satisfaction with Breasts domain. There is no overall or total score, only scores for each independent scale. All scales are transformed into scores ranging from 0-100. A higher score means greater satisfaction or better QOL
Change from baseline in WHO Disability Assessment Schedule V.2.0 after preoperative intervention and surgery, 6 weeks postoperative intervention, and after a three month observational period | Assessed at baseline (T0), within 1 week of completing the 2 weeks post-surgery (T1), within 1 week of completing the 6-weeks of postoperative exercise (T2), and within 1 week of completing the 3-months follow-up post-exercise (T3)
  Patient reported disability will be measured using the WHO Disability Assessment Schedule V.2.0 instrument. The scores assigned to each of the items are "none" (0), "mild" (1) "moderate" (2), "severe" (3) and "extreme" (4). These scores are summed for each item and are converted to a summary score ranging from 0 to 100 (where 0 = no disability; 100 = full disability).
Change from baseline in Shoulder pain and disability index (SPADI) after preoperative intervention and surgery, 6 weeks postoperative intervention, and after a three month observational period | Assessed at baseline (T0), within 1 week of completing the 2 weeks post-surgery (T1), within 1 week of completing the 6-weeks of postoperative exercise (T2), and within 1 week of completing the 3-months follow-up post-exercise (T3)
  Shoulder pain and disability will be measured using the 13 item SPADI assessing pain level and extent of difficulty with ADLs requiring the use of the upper extremities. The pain subscale has 5-items and the Disability subscale has 8-items. The pain scale is summed up to a total of 50 while the disability scale sums up to 80. The total SPADI score is expressed as a percentage where 0% indicates best and 100% indicates worst (i.e. a higher score shows more disability)
Change from baseline in Musculoskeletal Health Questionnaire (MSK-HQ) Schedule V.2.0 instrument after preoperative intervention and surgery, 6 weeks postoperative intervention, and after a three month observational period | Assessed at baseline (T0), within 1 week of completing the 2 weeks post-surgery (T1), within 1 week of completing the 6-weeks of postoperative exercise (T2), and within 1 week of completing the 3-months follow-up post-exercise (T3)
  Musculoskeletal joint, back, neck, bone and muscle symptoms such as aches, pains and/or stiffness will be assessed using the 14 item MSK-HQ. A summary score between 0-56 is computed; with a higher score indicating a better MSK-HQ status. There is also a question which asks patients to indicate, in the past week, how many days they have engaged in physical activity that has raised their heart rate for 30 minutes or more (0 to 7 days).
Change from baseline in 6 minute walk test (6MWT) after preoperative intervention and surgery, 6 weeks postoperative intervention, and after a three month observational period | Assessed at baseline (T0), within 1 week of completing the 2 weeks post-surgery (T1), within 1 week of completing the 6-weeks of postoperative exercise (T2), and within 1 week of completing the 3-months follow-up post-exercise (T3)
  To assess functional capacity, the investigators will record distance travelled, RPE, heart rate, estimated VO2max and oxygen saturation during a remotely supervised 6-minute walk test (6MWT), in accordance with ATS guidelines. The distance walked will be measured using manual tape measurement and validated using a cipher skin biosleeve
Change from baseline in 30 second chair to stand (30CST) after preoperative intervention and surgery, 6 weeks postoperative intervention, and after a three month observational period | Assessed at baseline (T0), within 1 week of completing the 2 weeks post-surgery (T1), within 1 week of completing the 6-weeks of postoperative exercise (T2), and within 1 week of completing the 3-months follow-up post-exercise (T3)
  To assess lower extremity strength and balance a remotely supervised 30 second chair to stand (30-CST) test will be performed. The number of times a patient comes to a full standing position from a chair will be recorded (the same chair will be used for all within-participant assessments).
Change from baseline in Hand Grip dynamometry after preoperative intervention and surgery, 6 weeks postoperative intervention, and after a three month observational period | Assessed at baseline (T0), within 1 week of completing the 2 weeks post-surgery (T1), within 1 week of completing the 6-weeks of postoperative exercise (T2), and within 1 week of completing the 3-months follow-up post-exercise (T3)
  Hand Grip dynamometry will be used as a measure of upper body muscular strength. The investigators will follow the Southampton protocol.
Change from baseline in Shoulder range of motion (RoM) after preoperative intervention and surgery, 6 weeks postoperative intervention, and after a three month observational period | Assessed at baseline (T0), within 1 week of completing the 2 weeks post-surgery (T1), within 1 week of completing the 6-weeks of postoperative exercise (T2), and within 1 week of completing the 3-months follow-up post-exercise (T3)
  To assess shoulder range of motion (RoM) the following movements will be performed under remote supervision; shoulder flexion, abduction, internal rotation, and external rotation. The RoM of each movement will be recorded using a cipher skin biosleeve and a single composite score, defined as the total of these four motions (sumRoM), calculated.
Change from baseline in Lymphedema after preoperative intervention and surgery, 6 weeks postoperative intervention, and after a three month observational period | Assessed at baseline (T0), within 1 week of completing the 2 weeks post-surgery (T1), within 1 week of completing the 6-weeks of postoperative exercise (T2), and within 1 week of completing the 3-months follow-up post-exercise (T3)
  Bilateral measurements will be made via a flexible tape with patients seated and their arm supported on a table with the shoulder in approximately 30° of forward flexion and 45° of elbow flexion. The investigators will use the landmarks method, where measurements will be taken at the wrist, elbow, and axilla plus two additional points either 10 cm distal to and proximal to the lateral epicondyle (Landmarks) or halfway between the wrist and elbow or elbow and axilla (Landmarks, Midpoint) (NLN position paper). Volumes will be then calculated by the sum of truncated cones (frustum) model for both Landmark and Landmark, Midpoint methods
Change from baseline in Habitual Physical Activity (active minutes) after preoperative intervention and surgery, 6 weeks postoperative intervention, and after a three month observational period | Assessed at baseline (T0), within 1 week of completing the 2 weeks post-surgery (T1), within 1 week of completing the 6-weeks of postoperative exercise (T2), and within 1 week of completing the 3-months follow-up post-exercise (T3)
  The investigators will track patient's habitual physical activity (i.e. outside of the prescribed exercise sessions) and sedentary behaviour via a Withings smartwatch (Steel HR) worn on patients left wrist (3 finger widths above the wrist bone). The Withings Steel HR is a high precision MEMS 3-axis accelerometer with heart rate infrared sense that provides estimates of time spent as 'active minutes'. The calculation of these minutes is based on Metabolic Equivalent of Task (METs)
Change from baseline in 4 day food diary after preoperative intervention and surgery, 6 weeks postoperative intervention, and after a three month observational period | Assessed at baseline (T0), within 1 week of completing the 2 weeks post-surgery (T1), within 1 week of completing the 6-weeks of postoperative exercise (T2), and within 1 week of completing the 3-months follow-up post-exercise (T3)
  Dietary intake will be assessed at each assessment point using a 4-day food diary.
Number of participants who experienced treatment-related adverse events (AEs) | Assessed 2 weeks post-surgery (T1), immediately after the 6-weeks of postoperative exercise (T2), and immediately after the 3 months follow up post exercise period (T3)
  Treatment-related adverse events (AEs) will be assessed via CTCAE and patient-reported outcomes CTCAE (PRO-CTCAE). Clinicians will report AEs at every consultation from T2 to T3. From the PRO-CTCAE, the investigators selected 12 core items including pain, fatigue, physical activity, bowel function, sleep, temperature, chill, sore mouth, and appetite (amscolme). The investigators will use an online reporting form that will ask patients to complete weekly for the 13 weeks between T2 and T3.
Chemotherapy completion rate | Assessed immediately after the 6-weeks of postoperative exercise (T2), and immediately after the 3 months follow up post exercise period (T3)
  For those patients who receive chemotherapy, chemotherapy completion rate will be assessed via relative dose intensity
Focus groups | Assessed immediately after the 6-weeks of postoperative exercise (T2), and immediately after the 3 months follow up post exercise period (T3)
  All participants will be invited to take part in a virtual focus group after completing the postoperative exercise intervention and at 3-months follow up to obtain qualitative data regarding topics such as patient preferences, intervention acceptability, and ideas for improving the intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Amtul Carmichael, Principal Investigator — University Hospitals of Derby and Burton NHS Foundation Trust
Locations (1):
- University Hospital Derby and Burton, Burton-on-Trent, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Data obtained through this study will be coded and made available via a publicly available repository (OSF: https://osf.io/v8azj/), with no protected health information included.
Supporting Information: Study Protocol
URL: https://osf.io/v8azj/